CLINICAL TRIAL: NCT00698048
Title: Serial Vasopressin and Copeptin Levels in Children With Sepsis and Septic Shock
Acronym: VaCoSS
Status: Completed | Type: Observational
Sponsor: Jan Hau Lee (Other Government)
Collaborators: National Medical Research Council (NMRC), Singapore (Other Government)
Responsible Party: Sponsor-Investigator, Jan Hau Lee, Dr Lee Jan Hau, KK Women's and Children's Hospital
Organization: KK Women's and Children's Hospital (Other Government)
Other Study IDs: NIG07nov002
Record Dates: First submitted 2008-06-12; First posted 2008-06-16 (Estimated); Last update posted 2015-09-09 (Estimated); Status verified 2015-09

CONDITIONS: Sepsis; Septic Shock
Keywords: Sepsis; Septic Shock; Vasopressin; Copeptin; Paediatrics
MeSH Terms: conditions — Sepsis; Shock, Septic; Diabetes Insipidus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: Controls
- 2: Sepsis
- 3: Septic Shock

SUMMARY:
Patients with severe infection can develop very low blood pressure. There are many mechanisms leading to this, and one of them appears to involve a hormone called vasopressin. In children as compared to adults, the mechanism and response to low blood pressure are different for reasons that are not clear. One possibility is the difference in the production and/or response to vasopressin. Vasopressin has become part of the treatment of children with low blood pressure in the setting of severe infection, when other treatment has failed, but its use is on the basis of animal and adult studies. The exact timing and dose is uncertain.

In this research study, the patients will receive standard treatment for sepsis and septic shock, and the investigators will measure the blood levels of vasopressin and a related compound called copeptin (both are required to understand the mechanism of control involved). Blood will need to be taken from patients without any sepsis so as to be able to compare the values in health and in sickness. The patient groups the investigators have chosen for this are those children who will have blood taken anyway as part of their routine care. The aim of this study is to develop an understanding of the body's hormonal response (with respect to vasopressin) to severe infection in children. The long-term aim is to improve the care of critically ill children with severe infection by using the most appropriate dose of vasopressin at the most appropriate time.

ELIGIBILITY:
Inclusion Criteria:

Control Group:

* Neonates admitted for neonatal jaundice requiring phototherapy
* Previously well patients admitted for elective gastrointestinal endoscopy, patients admitted for non-specific abdominal pain and
* Pre-operative patients for circumcision, inguinal hernias and chronic orthopaedic conditions

Study Group:

* The investigators will also enroll children with sepsis and septic shock
* Sepsis will be defined as proposed by the International pediatric sepsis consensus conference.
* Children will be recruited into the septic shock group if they have sepsis and features of cardiovascular organ dysfunction as defined by the same consensus conference.

Exclusion Criteria:

* Neonates weighing less than 2.5 kg
* Neonates less than 36 weeks gestation
* Children more than 16 years of age
* Patients with a history of congenital heart disease
* Patients with chronic renal impairment
* Patients with chronic liver impairment
* Patients on active chemotherapy
* Patients on chronic mineralocorticoids or glucocorticoids therapy
* Patients on long-term diuretic therapy
* Patients with central nervous system tumours
* Patients with developmental delay

Ages: 1 Day to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children between one day of age and sixteen years old.
Sampling Method: Non-Probability Sample
Enrollment: 136 (Actual)
Dates: Start 2008-08; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Vasopressin and copeptin levels | First 5 days of admission

CONTACTS AND LOCATIONS:
Overall Officials: Jan Hau Lee, MRCPCH(UK), Principal Investigator — KK Women's and Children's Hospital
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore